CLINICAL TRIAL: NCT02813915
Title: A Trial of a Non-Invasive Cardiac Output in Young Adults
Brief Title: Non-invasive Cardiac Output Monitor in Young Adults
Acronym: NICOM
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Cheetah Medical Inc. (Industry)
Responsible Party: Principal Investigator, Andrew Stasic, Associate Professor of Clinical Anesthesia, Indiana University
Other Study IDs: 1508764960
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Fluid Overload; Hypovolemia
Keywords: cardiac monitoring, Cheetah Medical, passive leg raises
MeSH Terms: conditions — Edema; Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Use of Cheetah medical NICOM: For those who consent to the study, the Cheetah NICOM will be used to obtain cardiac output, stroke volume, and fluid responsiveness.
  Interventions: Device: NICOM

INTERVENTIONS:
Device: NICOM — Use of NICOM and PLR to obtain patient fluid status

SUMMARY:
The investigators would like to study cardiac output, stroke volume, and fluid responsiveness on young adult pediatric patients undergoing anesthesia and surgery with the use of the NICOM, a non-invasive monitor. The NICOM method is non-invasive and provides reliable trending of cardiac output and stroke volume. Measuring cardiac output in conjunction with routine monitoring will provide a better assessment of intra-operative status.

DETAILED DESCRIPTION:
This study will involve measurements of cardiac output, stroke volume, and fluid responsiveness (change in stroke volume of ≥ 10%) obtained via passive leg raise (PLR) before and after anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* 18 -30 years of age
* presenting for surgery at Riley or University Hospital

Exclusion Criteria:

* younger than 18
* severely mentally handicapped
* orthopedic cases with leg injuries
* any other contraindications that would prevent or discourage passive leg raises
* if deemed ineligible by an investigator for any other reason.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients 18-30 years of age having surgery at Riley or University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-07-17; Primary Completion 2017-07-21 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Patient Fluid responsiveness | within 30 minutes post-anesthesia induction
  If patient is fluid responsive, Stroke Volume Index (SVI) will increase by 10% or greater compared to its baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Stasic, MD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: No